CLINICAL TRIAL: NCT06256445
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase Ⅲ Clinical Study to Evaluate Efficacy and Safety of AYP-101 for the Reduction of Submental Fat in Adults
Brief Title: Evaluate the Efficacy and Safety of AYP-101 for the Reduction of Submental Fat in Chin Area
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AMIpharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AYP-101-301
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Healthy
MeSH Terms: interventions — polyene phosphatidylcholine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AYP-101 (Experimental): 0.2 mL injections, 1.0 cm apart, up to 10.0 ml per treatment session at intervals of approximately 2 weeks for up to a maximum of 6 treatments
  Interventions: Drug: Polyene Phosphatidylcholine
- Placebo (Placebo Comparator): 0.2 mL injections, 1.0 cm apart, up to 10.0 ml per treatment session at intervals of approximately 2 weeks for up to a maximum of 6 treatments
  Interventions: Drug: Matching placebo of AYP-101

INTERVENTIONS:
Drug: Polyene Phosphatidylcholine — Formulated as an injectable solution containing Polyene Phosphatidylcholine at concentration of 25 mg/mL
  Other Names: AYP-101
  Arms: AYP-101
Drug: Matching placebo of AYP-101 — Phosphate buffered saline placebo for injection
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
To Evaluate Efficacy and Safety of AYP-101 S.C injection for the Reduction of Submental Fat in Adults

DETAILED DESCRIPTION:
This study is to evaluate efficacy and safety of AYP-101 S.C injection for the reduction of Submental Fat who wish improvement in the appearance of moderate to severe convexity or fullness associated with Submental Fat in adults

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 19 to 65 (inclusive)
2. Patient with submental subcutaneous fat deposited who meet all of the following:

   * Patient with ER-SMFRS and SR-SMFRS Grade 2 (moderate) or 3 (severe) at visit 1
   * Subject Self Satisfaction Scale (SSSS) Grade 2 (slightly dissatisfied) or less at visit 1
3. Patient who has stably maintained body weight for the past 6 months (weight change within ±10% of subject's weight); agrees to refrain from exercise and diet that may affect the study result during the study period and maintain pre-study exercise/diet during the study period
4. Able to comply with the protocol visit schedule and plans
5. Voluntarily provides written informed consent

Exclusion Criteria:

1. Allergic to IP component (soy) and lidocaine or medical devices used in this clinical trial (sterile permanent marker, alcohol swab, administration site design grid pad, injection needle, etc.)
2. Has morbid obesity of central, endocrine, and genetic nature (BMI ≥ 35 kg/m2 at screening)
3. History of plastic surgery (liposuction) or injection containing phosphatidylcholine or deoxycholic acid at the planned IP administration site for the purpose of submental fat reduction or history of double jaw surgery
4. History of following procedures at the planned IP administration site

   * Thread lifting, implants, dermal fillers with active ingredient other than hyaluronic acid or collagen, or semi-permanent fillers within 12 months prior to visit 2
   * Dermal fillers with active ingredient hyaluronic acid or collagen or Botulinum toxin procedure within 6 months prior to visit 2 (including entire chin and neck area)
   * Focused ultrasound, radiofrequency or cryolipolysis within 6 months prior to visit 2
   * Laser therapy, optic therapy, or chemical dermabrasion procedure within 3 months prior to visit 2
5. Deemed inappropriate for the study by the investigator, such as the following:

   * Skin at the administration site is sagging or deformed
   * Has a prominent platysmal band under the chin
   * Has a short chin; jawbone in the lower jaw developed less than normal
   * Has a condition (e.g., cervical lymphadenopathy), inflammation, wound or surgical scar in the chin or the neck that is deemed to affect study assessments
   * Has any other factors deemed to affect evaluations by the investigator (evaluator)
6. History of dysphagia or current symptoms of dysphasia
7. Diagnosis of heart disease (heart failure, unstable angina, myocardial infarction) or brain disease (stroke, cerebral hemorrhage, cerebral infarct) within 6 months of screening
8. Has a condition during this study period that requires medication with NSAIDs (arthritis, lung diseases, etc.)
9. Uncontrolled hypertension (sitSBP ≥180 mmHg or sitDBP ≥110 mmHg at screening)
10. Uncontrolled type 2 diabetes (HbA1c > 9% at screening) or type 1 diabetes
11. Has an autoimmune disease or receiving immunosuppressants
12. Receiving anticoagulants such as warfarin and clopidogrel or has a coagulation disorder
13. Has thyromegaly or hyperthyroidism
14. HIV-positive
15. Diagnosis of malignancy within the last 5 years
16. Severe renal dysfunction (serum creatinine > 2.0 mg/dl at screening)
17. Severe liver dysfunction (ALT, AST or ALP > upper limit of normal x 2.5 at screening)
18. A history of or currently suffering from a serious psychiatric condition (e.g., depression, schizophrenia, epilepsy, alcoholism, drug addiction, anorexia, bulimia)
19. Administration of drugs that may affect the body weight and lipid metabolism, such as appetite suppressants, oral steroids, thyroid hormones, amphetamines, cyproheptadine, phenothiazines or drugs that may affect absorption, metabolism and excretion within 3 months of screening
20. Receipt of any other IPs within 3 months prior to IP administration
21. Pregnant or lactating women, or subjects who are planning to become pregnant
22. Failure to agree to use a contraceptive method that is highly effective when used correctly, alone or in combination, continuously throughout the study and up to 3 months after the final IP administration
23. Deemed ineligible to be a study subject by the investigator

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Co-primary Outcome Measure 1 | at 12 weeks after the final administration compared to baseline
  Ratio of subjects with at least 1 grade improvement in both ER-SMFRS(Evaluator Reported Submental Fat Rating Scale) and SR-SMFRS(Subject Reported Submental Fat Rating Scale)
Co-primary Outcome Measure 2 | at 12 weeks after the final administration compared to baseline
  Ratio of subjects with at least 2 grades improvement in both ER-SMFRS and SR-SMFRS

SECONDARY OUTCOMES:
At least 1 grade improvement in both ER-SMFRS and SR-SMFRS | at 4 weeks after the final administration compared to baseline
  Ratio of subjects with at least 1 grade improvement in both ER-SMFRS and SR-SMFRS
At least 2 grade improvement in both ER-SMFRS and SR-SMFRS | at 4 weeks after the final administration compared to baseline
  Ratio of subjects with at least 2 grades improvement in both ER-SMFRS and SR-SMFRS
At least 1 grade improvement in ER-SMFRS | at 4 and 12 weeks after the final administration compared to baseline
  Ratio of subjects with at least 1 grade improvement in ER-SMFRS
At least 2 grades improvement in ER-SMFRS | at 4 and 12 weeks after the final administration compared to baseline
  Ratio of subjects with at least 2 grades improvement in ER-SMFRS
At least 1 grade improvement in SR-SMFRS | at 4 and 12 weeks after the final administration compared to baseline
  Ratio of subjects with at least 1 grade improvement in SR-SMFRS
At least 2 grades improvement in SR-SMFRS | at 4 and 12 weeks after the final administration compared to baseline
  Ratio of subjects with at least 2 grades improvement in SR-SMFRS
SSSS(Subject Self Satisfaction Scale) | at 4 and 12 weeks after the final administration
  Ratio of subjects with SSSS of at least 4 points
PR-SMFIS(Patient Reported Submental Fat Impact Scale) | at 4 and 12 weeks after the final administration
  Change in average PR-SMFIS score from baseline, In detail, it is a tool on which subjects measure how their submental fat looks on a scale of 0 to 10 points b y responding to 6 questions.
  Item 1 is in regard to satisfaction, and items 2 to 6 are questions in regard to dissatisfaction; all items will be calculated on a dissatisfaction scale* and mean will be calculated.
  * Item 1 dissatisfaction scale = 10 (points) - Item 1 score
  * Items 2 to 6 dissatisfaction scale = each item score
  Each item in the PR-SMFIS is scored from 0 to 10, with a higher total score indicating greater dissatisfaction.
PGIC(Patient Global Impression of Change) | at 4 and 12 weeks after the final administration
  PGIC evaluation
3D imaging | at 4 and 12 weeks after the final administration
  Change in subject's submental fat volume by 3D imaging from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Beomjoon Kim, MD, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- Chung-Ang University Hosptial, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No